CLINICAL TRIAL: NCT02258165
Title: Impact of Gated PET/CT on the Diagnosis of Distant Metastases of Advanced Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Impact of Gated PET/CT in the Diagnosis of Advanced Ovarian Cancer
Acronym: IMAGE
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: The University of Queensland (Other); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMAGE
Record Dates: First submitted 2014-09-08; First posted 2014-10-07 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Cancer Stage III; Ovarian Cancer Stage IV
Keywords: ovarian cancer; imaging; gated PET/CT scan
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced ovarian cancer: gated PET/CT imaging
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — PET/CT (without respiratory gating) is performed on an ad-hoc basis in patients with advanced ovarian cancer in the lead up to surgery. The sensitivity of PET/CT for detecting low volume pleural disease is likely reduced by respiratory motion during the ten minute acquisition time over the chest. By "freezing" this respiratory motion with respiratory gating, we hope that gated PET/CT detection of pleural metastases will improve over non-gated PET images.

SUMMARY:
This study will be the first prospective study enrolling consecutive patients with advanced ovarian cancer to determine the prevalence of thoracic and extra-abdominal involvement in this patient group and the relative value of gated PET and CT for diagnosing extra-abdominal involvement. This study will also answer a number of other stil unanswered questions: the impact of gating and the impact of gated PET on clinical management of patients with advanced ovarian cancer. This study also individualises patients' treatment to allow patients who may benefit most form optimal surgical cytoreduction and those who are better treated by neoadjuvant

DETAILED DESCRIPTION:
This study directly compares standard CT scanning with PET/CT scanning with gating (computer adjusted for breathing excursions) in patients with advanced EOC. The primary objective of this study is to obtain definitive evidence on the value of gated PET/CT compared to current standard imaging (CT scan) for the diagnosis of extra-abdominal and thoracic involvement. This study will give precise estimates on the sensitivity and specificity of CT compared with gated PET/CT, and allow calculation of the positive predictive value and negative predictive value. The proportion of patients upstaged to Stage IV (extra-abdominal involvement) from Stage III by gated PET/CT will be calculated.

Secondary objectives are to establish:

* The impact of gated PET/CT images on clinical management (changes to planned treatment; detection of metastatic spread to "unexpected" sites).
* The validity of gated PET/CT positive (FDG avid) findings through histological evaluation.
* We will also receive information of "unusual" (unexpected) FDG positive metastatic lesions that would normally not noticed on CT scans.

Current standard treatment for patients with advanced EOC is upfront surgery as long as all tumour is confined to the pelvis and the abdomen. Unfortunately, EOC is often found at distant sites where it was not suspected during surgery (which is too late). If the surgeon had had prior knowledge of this disease distribution, the surgeon would not have subjected the patient to a long and invasive surgical procedure. Instead they but would have referred the patient to upfront chemotherapy, which is widely accepted clinical practice throughout Australia.

This study aims to increase the diagnostic accuracy of preoperative medical imaging and subject a larger group of patients with advanced EOC to accurate management.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥18 years of age
* Suspected or histologically/cytologically proven Stage III or IV epithelial ovarian, fallopian tube, and primary peritoneal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤3
* Negative serum or urine pregnancy test in pre-menopausal women and women < 2 years after the onset of menopause
* Signed written informed consent

Exclusion Criteria:

* Estimated life expectancy of <6 months
* Recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Laparotomy performed as component of staging/clinical management prior to gated PET/CT being performed.
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with advanced ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients upstaged from Stage IV from Stage III by gated PET/CT | one to six months
  The primary hypothesis is that the true prevalence of extra-abdominal involvement diagnosed by gated PET/CT will be higher than the prevalence deteted by CT.

SECONDARY OUTCOMES:
Impact of gated PET/CT images on clinical management | one to six months
  Changes to planned treatment for ovarian cancer based on the detection of metastatic spead to "unexpected sites"
The validity of gated PET/CT positive (FDG avid) findings through histological evaluation | one to six months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Study Chair — Queensland Centre for Gynaecological Cancer
Locations (2):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Virili F, Obermair A, Sanjida S, Nicklin JL, Garrett A, Land R, Tang A, Campbell L, Gebski V, Thomas P. Impact of gated FDG PET/CT on the staging of patients with suspected or proven newly diagnosed advanced epithelial ovarian, fallopian tube, and primary peritoneal cancer: results from a non-randomized, phase II clinical trial. Int J Gynecol Cancer. 2025 Jan 6:ijgc-2024-005633. doi: 10.1136/ijgc-2024-005633. Online ahead of print. PMID 39237158